CLINICAL TRIAL: NCT05794880
Title: Matched Unrelated Donor and Partially Matched Related Donor Peripheral Stem Cell Transplantation With Alpha/Beta T-Cell and B-Cell Depletion for Patients With Hematologic Malignancies With Targeted ATG Dosing Pilot Study, IDE 13641
Brief Title: MCW Alpha/Beta T-Cell and B-Cell Depletion With Targeted ATG Dosing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Amy Moskop, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-MOSKOP-MABD
Record Dates: First submitted 2023-03-08; First posted 2023-04-03 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Leukemia; Acute Myeloid Leukemia in Remission; Myelodysplasia; Acute Lymphoblastic Leukemia in Remission; Chronic Myelogenous Leukemia - Chronic Phase; Chronic Myelogenous Leukemia, Accelerated Phase; Chronic Myelogenous Leukemia With Crisis of Blast Cells; Biphenotypic Acute Leukemia; Lymphoblastic Lymphoma; Burkitt Lymphoma; Burkitt Leukemia; Lymphoma After Relapse; Other Malignant Hematologic Diseases in Remission
MeSH Terms: conditions — Leukemia; Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Alpha/Beta T cell depletion (TCD) plus CD19+ depletion (Experimental): Alpha beta T cell and B cell depleted allogeneic transplantation with individualized dosing of ATG for patients with hematologic malignancies
  Interventions: Device: Magnetic-Activated Cell Sorter (CliniMACS, Miltenyi)

INTERVENTIONS:
Device: Magnetic-Activated Cell Sorter (CliniMACS, Miltenyi) — Participants in this study will receive a blood stem cell transplant, which will use an investigational device called the CliniMACs device to remove alpha/beta T cells and B cells from the blood cells collected from the donor. This is called T cell depletion and B cell depletion.

SUMMARY:
This is a single arm pilot study for patients with hematologic malignancies receiving unrelated or haploidentical related mobilized peripheral stem cells (PSCs) using the CliniMACS system for alpha/beta T cell depletion plus CD19+ B cell depletion with individualized ALC-based dosing of ATG to study impact on engraftment, GVHD, and disease free survival

ELIGIBILITY:
Inclusion Criteria:

1. Patient age < 25 years. Both genders and all races eligible.
2. Disease eligibility

   * Acute myeloid leukemia, primary or secondary - Disease status: MRD negative (flow MRD ≤ 0.1%)
   * Myelodysplasia
   * Acute lymphoblastic leukemia - Disease status: MRD negative
   * Chronic myelogenous leukemia - Disease status: chronic phase, accelerated phase or blast crisis now in second chronic phase
   * Mixed lineage or biphenotypic acute leukemia- Disease status: MRD negative
   * Lymphoblastic lymphoma - Disease status: in remission
   * Burkitt's lymphoma/leukemia - Disease status: in remission
   * Lymphoma after relapse - Disease status: in remission
   * Other malignant hematologic diseases in remission (to be approved by PI)
3. Karnofsky Performance Status ≥ 60% for patients 16 years and older and Lansky Play Score ≥ 60 for patients under 16 years of age (Appendix 1)
4. Evaluation of organ status as per MCW BMT SOP
5. Infectious disease criteria: No active untreated infection. Patients with possible fungal infections must have had at least 2 weeks of appropriate anti-fungal antibiotics and be asymptomatic.
6. Signed consent by parent/guardian or able to give consent if ≥18 years.
7. Negative pregnancy test for patients capable of childbearing potential
8. Sexually active patients capable of child-bearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment. Sexually active men must agree to use barrier contraceptive for the duration of treatment.

Donor Eligibility:

1. Unrelated donor meets National Marrow Donor Program criteria for donation
2. Infectious disease testing
3. MCW BMT procedures apply for determining donor eligibility, including donor screening and testing for relevant communicable disease agents and diseases.
4. Only Peripheral blood stem cells will be used for stem cell source on this study therefore donor must be willing to undergo G-CSF mobilization and stem cell apheresis. Donor matching. High resolution typing at all loci to be performed.
5. Unrelated Donor:

   a. HLA typing of at least 10 alleles is required. Donor must be matched at 9/10 or 10/10 alleles (HLA A, B, C, DRB1, DQB1).Donor and collection center willing to undergo mobilization and apheresis
6. Haploidentical Related Donor:

   1. Haploidentical parent or other related donor: Minimum match level full haploidentical (at least 5/10; HLA A, B, C, DRB1, DQB1 alleles), but use of haploidentical donors with extra matches (e.g. 6, 7, or 8/10) encouraged.

Exclusion Criteria:

1. Patients who do not meet disease, organ, or infectious criteria.
2. No suitable donor
3. Pregnant or lactating patients are ineligible as many of the medications used in this protocol could be harmful to unborn children and infants
4. Receiving concomitant chemotherapy, radiation therapy; immunotherapy or other anti-cancer therapy for treatment of disease other than is specified in the protocol. Maintenance or other post-HCT therapy can be considered after discussion with the study PI.
5. Participating in a concomitant Phase 1 or 2 study involving treatment of disease
6. Active malignancy other than eligible disease specified in the protocol. Patients with prior malignancy can be eligible as long as at least 1 year post treatment for that malignancy.

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate incidence and extent of aGVHD and engraftment in patients receiving alpha/beta T cell depleted and CD19+ B cell depleted stem cell transplant with individualized ALC-based dosing of ATG | 1 year

SECONDARY OUTCOMES:
Evaluate incidence of chronic GVHD | 5 years
Evaluate time to platelet engraftment | 1 years
Assess incidence of viral infections | 2 years
Evaluate incidence of relapse/progressive disease | 2 years
Evaluate incidence of treatment-related mortality (TRM). | 2 years
Evaluate overall and relapse free survival (RFS) at 1 year | 1 years

OTHER OUTCOMES:
Assess tempo of CD4+ T cell reconstitution. | 2 years
Assess tempo of immune reconstitution. | 2 years
Assess ATG exposure using pre- and post- HCT AUC estimates using ATG dosing module | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No